CLINICAL TRIAL: NCT03139877
Title: Pediatric Obesity Observational Prospective Trial: Microbiome and Metabolism During Obesity Target Therapeutics
Brief Title: Pediatric Obesity Observational Prospective Trial
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00074729
Record Dates: First submitted 2017-03-15; First posted 2017-05-04 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples: Samples will be kept at 4ºC for < 18 hours prior to moving to the lab -80ºC freezer.
  Using the Human Microbiome Roadmap (REFS), Ribosomal DNA will be amplified using multiplexing primers per Caparoso et al method. Pooled amplicons will be sequenced. Sequences will be stored on the Center for Genomes in Microbial Systems (GeMS) without PHI.
  A 20 mL(milliliter) blood sample will be collected for isolation of mononuclear cells and plasma for genetic and metabolomics studies.
  Sampling will not exceed 2 ml/kg or 90 ml over the course of the study. Mononuclear cell DNA will be isolated from peripheral samples and applied to a focused polymorphism analysis for 29 obesity risk alleles using Sequenom technology at the David H. Murdock Research Institute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HLP: Intervention Cohorts:The intended target population is the adolescent with a BMI ≥ 95th percentile.
  Healthy Lifestyles Program(HLP) will serve as the primary recruitment site for the intervention cohort. A prospective, longitudinal observational case control study will be performed. All participants will receive HLP standard of care (intensive lifestyle modification and access to Bull City Fit.) Groups: (1) HL-only, (2) HL + Low carbohydrate diet, (3) HL + weight loss medication(s) and (4) HL + Bariatric surgery.
  Participants will be assigned to groups as per usual HLP clinical care, based on established standards and guidelines, expert medical provider recommendations, and family preference.
- Healthy Weight Siblings: Healthy weight siblings of HLP participants who meet age and BMI criteria will be offered enrollment at the time their overweight sibling is consented to provide comparative data. This group will be asked to provide a fecal and blood sample at one time point.
- Healthy Weight age/sex matched controls: Healthy weight, age and gender matched patients will be recruited from the Duke Children's primary care practice Participants will be recruited at the time of their annual physical to provide comparative data.
  This group will be asked to provide a fecal and blood sample at one time point.

SUMMARY:
Using an observational case-control cohort design, the investigator aims to define the mechanisms underlying microbiome regulation of metabolism in adolescence before and after medically indicated therapies for obesity. The investigator's overarching hypothesis is that gut bacteria control host weight, insulin sensitivity, and response to weight-loss treatments by modifying host metabolism.

DETAILED DESCRIPTION:
Intervention Cohorts: A prospective, longitudinal observational case control study will be performed. All subjects will receive Healthy Lifestyle Program (HLP) standard of care, which includes intensive lifestyle modification and free participation in Bull City Fit. Four groups of participants receiving obesity treatment will be enrolled: (1) HLP-only, (2) HLP + Low carbohydrate diet, (3) HLP + weight loss medication(s) and (4) HLP + Bariatric surgery. Consistent with the observational design of this study, study participants will be assigned to each group as per usual HLP clinical care, based on established standards and guidelines, expert medical provider recommendations, and family preference.

Comparison Cohort: two comparison groups be enrolled:(1c) healthy siblings of enrolled intervention subjects and (2c) age/sex matched controls recruited from the Duke Children's Primary Care Clinic.

Up to 350 participants will be enrolled, with the goal of 295 evaluable participant data. The study period is six months for all groups with the exception of the bariatric surgery group which will last from baseline until after surgery, up to 12 months. The comparison groups will have one visit at baseline only.

Stool Sample Collection: Participants in both intervention and comparison groups will provide a fecal sample at enrollment or within 3 days of enrollment. Participants in intervention groups (Groups 1-4) will provide additional fecal samples at 1.5, 3, 4.5, and 6 months. Given that the ability to collect fecal samples is unpredictable, the investigator will develop a standard operating procedure along the following guidelines:

1. At the first visit, if the subject cannot provide a sample at the time of enrollment, the investigator will give the participant/parent a cooler/ice pack and sample collection kit. The investigator will ask the subject to provide the "baseline" sample within 3 days of the first visit. The sample will be refrigerated for up to 24 hours prior to pick up by the clinical research staff or delivery by the parent/guardian, with compensation for miles. With pick up or delivery a new cooler and freezer pack as well as sample collection kit will be provided for the following sample collection.
2. Within a 2-week window, centered on collection points 1.5 and 4.5 months, the subjects will provide additional samples. They may either have the samples picked up within 24 hours of collection (with refrigeration from collection to pick up) or get reimbursed for mileage.
3. For the 3-month and 6-month collections, which occur in conjunction with a regularly scheduled Healthy Lifestyles visit, the patients will collect a sample within 24 hours prior to the visit and bring with them to clinic. At the 3-month visit they will be sent home with new collection kits, freezer packs, and coolers.
4. If a patient cannot provide a sample within 24 hours of a clinic visit or a sample is missed, we will still collect a sample as soon as the patient is able to provide it and arrange for pickup or delivery as outlined below, noting the sample as "out of window."

Plasma sample collection: Participants in intervention groups will provide a 20mL blood samples at baseline, 3 and 6 months at the time of a regular HLP visit. The standard HLP clinical protocol is to draw fasting labs at baseline and 6 months, so no additional blood draws beyond what is required for clinical care will be required at those visits. However, HLP patients do not typically have a blood draw at 3 months, so participants will be asked for a blood sample at 3 months they would not otherwise require. Participants in comparison groups (Groups 1c, 2c) will be asked for a blood sample at enrollment only; they would not otherwise require this sample.

Analysis of samples: Fecal samples will be analyzed for the composition of the microbiota using DNA sequencing methods. Specific bacteria associated with obesity will be isolated from fecal samples and studied in the laboratory for their metabolism. A subset of fecal samples will be transferred into the intestinal tracts of germ free mice to study the effects on their metabolism. Participant plasma will be analyzed for panels of metabolites that are associated with diabetes mellitus and obesity. Blood mononuclear cell DNA will be used for focused genetic testing to identify genetic changes associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 10-18 years
* Sexual Maturity Rating 2 or above (pubertal)
* Age- and gender-specific BMI ≥ 95th percentile
* Expected enrollment in Healthy Lifestyles Clinical Program > 6 months

Exclusion Criteria:

* Antibiotic use in the 1 month prior to expected enrollment
* Anticipated antibiotic use during the course of the study.
* Immunodeficiency or prior transplantation
* Type 1 diabetes mellitus
* Inborn error of metabolism
* No fluency in English or Spanish
* Identifiable cause of obesity including hypothyroidism, Cushing syndrome, known genetic obesity syndrome including melanocortin receptor 4 mutation, drug-induced obesity including steroids or anti-psychotics
* Significant medical or mental health condition that precludes treatment
* Receiving insulin
* Plans to move away from area in next 6 months
* Weight loss of >5% total body weight in prior 3 months
* Pregnancy (self-report, confirm with noted last menstrual period in chart)
* Home outside of a 50 mile radius from the HL Clinic.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Duke Healthy Lifestyles (HL) Clinic Patients with BMI>95%
  1. c) Normal-weight siblings of patients presenting to the Duke Healthy Lifestyles Clinic
  2. c) Normal weight age/sex-matched controls presenting for well-child care to Duke Children's Primary Care clinic
Sampling Method: Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (kg/m2) | Baseline and 6 months
  We will measure weight (in kilograms) and height (in cm) for all subjects at baseline and at 6 months (12 months for the surgery group). The between-group difference in Body Mass Index change will be reported.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and 6 months
  Blood pressure will be measured at baseline and 6-months (12-months for the surgery group) using standard methods, and change in blood pressure between groups will be reported
Change in cardiovascular fitness | Baseline and 6 months
  We will perform a 3-minute standardized stepping test at baseline and 6-months (12 months for surgery group) and compare between-group differences in heart rate change with step test.
Change in fasting blood cholesterol | Baseline and 6 months
  We will measure fasting blood cholesterol at baseline and at 6-months (12 months for surgery group) and compare between-group differences in total cholesterol.
Change in fasting blood glucose | Baseline and 6 months
  We will measure fasting blood glucose at baseline and at 6-months (12 months for surgery group) and compare between-group differences in fasting blood glucose.
Change in stool microbiota profile | Baseline and every 6 weeks up to 6 months (0m, 1.5m, 3m, 4.5m, 6m)
  Fecal samples will be analyzed for the composition of the microbiota by extracting and sequencing the RNA from the organisms. We will report the communities of microbes at each time point.
Change in blood metabolites | Baseline, 3 months and 6 months
  Blood samples will be analyzed for a panel of metabolites that may be produced by the intestinal microbiota. We will report the metabolic profiles at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCann JR, Yang C, Bihlmeyer NA, Tang R, Truong T, An J, Jawahar J, Ilkayeva O, Muehlbauer MJ, Hu Z, Dressman HK, Poppe L, Granek JA, David LA, Shi P, Balikcioglu PG, Shah SH, Armstrong SC, Newgard CB, Seed PC, Rawls JF. Branched chain amino acid metabolism and microbiome in adolescents with obesity during weight loss therapy. medRxiv [Preprint]. 2025 Jun 9:2025.02.03.25321363. doi: 10.1101/2025.02.03.25321363. PMID 39974080
- [Derived] Suarez L, Skinner AC, Truong T, McCann JR, Rawls JF, Seed PC, Armstrong SC. Advanced Obesity Treatment Selection among Adolescents in a Pediatric Weight Management Program. Child Obes. 2022 Jun;18(4):237-245. doi: 10.1089/chi.2021.0190. Epub 2021 Nov 9. PMID 34757829